CLINICAL TRIAL: NCT05220956
Title: Impact of Time-restricted Feeding on Hepatic Steatosis in NAFLD
Brief Title: Impact of Time-restricted Feeding in NAFLD
Acronym: NAFLD-TRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jörn M. Schattenberg, Prof. Dr. Jörn M. Schattenberg, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 21-00784
Record Dates: First submitted 2021-06-22; First posted 2022-02-02 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Fatty Liver Disease; Fatty Liver; Fatty Liver, Nonalcoholic
Keywords: liver fibrosis; time restricted feeding
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Liver Cirrhosis; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled study with NAFLD-patients. One arm will undergo a TRF diet (Time-Restricted Feeding) for 12 weeks. The control arm is not subject to any time restrictions concerning eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (Other): This arm will undergo a TRF diet (Time-Restricted Feeding) for 12 weeks.
  Interventions: Behavioral: Intermittent fasting
- DGE diet (Other): This control arm is not a subject to any time restrictions concerning eating, solely patients will be trained according to the 10 rules of healthy nutrition of the DGE.
  Interventions: Behavioral: DGE diet

INTERVENTIONS:
Behavioral: Intermittent fasting — One arm will undergo a TRF diet (Time-Restricted Feeding) for 12 weeks while both arms undergo a training according to the 10 rules of healthy nutrition of the DGE.
  Other Names: Time restricted feeding
  Arms: Intermittent fasting
Behavioral: DGE diet — The control arm is not a subject to any time restrictions concerning eating while both arms undergo a training according to the 10 rules of healthy nutrition of the DGE.
  Arms: DGE diet

SUMMARY:
This is a randomised controlled study of patients with Non-Alcoholic Fatty Liver Disease (NAFLD).

Patients will be trained according to the 10 rules of a healthy nutrition according to the German Association for Nutrition (DGE).

One arm will undergo Time-Restricted Feeding (TRF) for 12 weeks. The control arm is not subject to any time restrictions concerning eating.

It will be investigated whether TRF improves insulin sensitivity, impacts on metabolic inflammation and reduces liver steatosis.

DETAILED DESCRIPTION:
Patients are recruited in the Liver Outpatient Clinic of the University Medical Center of Mainz.

About 100 patients will be enrolled in this pilot study. Inclusions criteria are exclusions of known causes of liver injury, Body Mass Index (BMI) > 25 kg/m^2, severe steatosis according to CAP ≥ 300 dB/m and absence of advanced fibrosis according to liver stiffness < 13 kPa.

Following the written consent, all patients will be trained to undertake a 2-week lead-in period of DGE.

Beginning in week 3 (Visit 2), an interventional group and a control group are generated through randomisation. The interventional group is instructed to follow TRF, whereas the control group is not subject to any time restrictions. Both arms will be accompanied for a duration of 12 weeks.TRF diet is based on temporal food consumption between 8:00 a.m. and 16:00 p.m., thus a 16 hour lasting period. After 10 weeks from the completion of the experimental phase (wash-out period), there will be the "end of follow up" visit.

The whole duration of the study is 24 weeks (2 weeks lead-in, 12 weeks intervention and 10 weeks post-intervention investigation).

Transient elastography (Fibroscan) is conducted at the screening visit, randomization visit, and at weeks 8, end of treatment visit and end of study visit. Spleen stiffness measurement is performed at randomization visit, week 8 and end of treatment visit. There will be 5 visits at the study center (screening, randomization, week 8, end of treatment and end of study) and 2 phone visits (week 6 and week 12). At each visit clinical events, body weight and standard laboratory parameters, identification of the CAP and stiffness values will be collected. Participants will fill in questionnaires capturing quality of life. At randomization visit and end of treatment visit, an OGTT will be performed to assess insulin sensitivity.

Adverse events will be recorded. Phone visits are used to survey the safety of patients.

Non-adherence to TRF for 2 days per week (20% of the total study period) has been selected as cut off to define treatment failure at per-protocol analysis.

ELIGIBILITY:
Patients with steady medication during the last 3 months. A diabetes mellitus must not be decompensated (HbA1c <6.5%). Patients with advanced fibrosis - defined about the non-invasive Fibroscan-procedure (Fibroscan >13 kPa) - will not be included.

Complete inclusion criteria:

1. Age between 18 and 75 years
2. Body Mass Index (BMI) > 25 kg/m2
3. Grade 3 steatosis evaluated by with CAP ≥ 300 dB/m and exclusion of known causes of liver steatosis
4. Liver elastography < 13 kPa
5. Capability to understand the study and the individual consequences of participation
6. Signed and dated declaration of agreement in the forefront of the study

Complete exclusion criteria:

1. Liver cirrhosis
2. Hepatocellular carcinoma or non-curative treated carcinoma
3. Alcohol consumption >20g (female) und >30 g (male)/day
4. Other causes of chronic liver disease (HBV, HCV, HDV, HEV, HIV), autoimmune diseases or chronic cholestatic liver disease, hereditary haemochromatosis, Wilson disease, α-1-Antitrypsin deficiency
5. Medications which cause liver disease or secondary NAFLD (e. g. Tamoxifen, systemic Corticosteroids, Methotrexate, Tetracycline, Estrogens, Valproic acid)
6. Changes in body weight > 5% in the last 6 months
7. Statins and/ or other fat-reducer medications if not taken in steady dosage during at least 4 weeks
8. Uncontrolled diabetes type 2 defined as HbA1c value > 9.0% or insulin depending type 2 diabetes
9. Pregnancy
10. Immunologic or inflammatory disease (e. h. systemic lupus erythematodes)
11. Patients after organ transplantations
12. Missing or lacking consent capability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of TRF on liver steatosis by CAP (dB/m) | 12 weeks
  The primary outcome of interest is a change in CAP value of a least 20 db/m with TRF

SECONDARY OUTCOMES:
Changes in liver fibrosis by liver stiffness (kPa) under TRF | 12 weeks
  Liver elastography performed as surrogate marker of liver fibrosis
Changes in FIB-4 as indirect non-invasive tools of liver fibrosis | 12 weeks
  Changes in the surrogate marker of liver fibrosis FIB-4
Evaluation of changes in direct non-invasive tool of liver fibrosis ELF | 12 weeks
  Performed as surrogate markers of liver fibrosis
Evaluation of changes in direct marker of liver fibrogenesis PRO-C3 (ng/ml) | 12 weeks
  Performed as surrogate markers of liver fibrosis
Evaluation of changes in liver-specific quality of life | 12 weeks
  Evaluation of Patient Reported Outcomes using the Chronic Liver Disease Questionnaire (CLDQ). The CLDQ uses 29 items in four domains, each scored on a Likert scale from 1 (all of the time) to 7 (none of the time) representing the frequency of clinical symptoms and emotional problems in the last two weeks. Results are reported in the six subscale scores (abdominal symptoms, fatigue, systemic symptoms, activity, emotional functioning, worry) and a CLDQ overall score.
Evaluation of changes in insulin sensitivity | 12 weeks
  Changes in insulin sensitivity by indexes derived by HOMA-IR score
Evaluation of changes in the gut microbiota | 12 weeks
  Evaluation of 16S rRNA gene sequencing for species and strain-level microbiome analysis.
Evaluation of changes in markers of oxidative stress (AGEs) | 12 weeks
  AGEs as surrogate markers of oxidative stress
Changes in spleen volume by spleen stiffness under TRF | 12 weeks
  Spleen stiffness performed as surrogate of spleen volume

CONTACTS AND LOCATIONS:
Overall Officials: Jörn M. Schattenberg, Prof., Principal Investigator — 1. Medical Department
Locations (1):
- University Medical Center of the Johannes Gutenberg Univeristy, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No
The transfer of data to third parties including publication will be exclusively in form of double pseudo-anonymized data, i.e. cannot be assigned to a person.